CLINICAL TRIAL: NCT05030571
Title: The Effects of Double Plasma Molecular Adsorption System in Acute on Chronic Liver Failure Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB.216/64
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Acute-On-Chronic Liver Failure; Acute on Chronic Hepatic Failure
Keywords: Hemoperfusion; Acute-On-Chronic Liver Failure; Cytokine adsorbant therapy; HA-330
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive DPMAS extracorporeal treatment one session per day for 3 consecutive days plus standard therapy. We plan to use blood flow rate of 100-120 ml/hour with filtration fraction for plasma separation of 25-30%. DPMAS circuit consist of Plasmaflo OP cartridge (Asahi Medical, Tokyo, Japan), Ion exchange resin hemoperfusion cartridge (BS330; Jafron, Zhuhai City, China), and Neutral adsorption resin hemoperfusion cartridge (HA330-II; Jafron, Zhuhai City, China) We do not use any anticoagulant.
  Interventions: Device: DPMAS; Other: standard treatment
- Standard care (Active Comparator): Standard treatment according to EASL Clinical Practical Guidelines on the management of acute (fulminant) liver failure 2017
  Interventions: Other: standard treatment

INTERVENTIONS:
Device: DPMAS — DPMAS circuit consist of Plasmaflo OP cartridge (Asahi Medical, Tokyo, Japan), Ion exchange resin hemoperfusion cartridge (BS330; Jafron, Zhuhai City, China), and Neutral adsorption resin hemoperfusion cartridge (HA330-II; Jafron, Zhuhai City, China)
  Arms: Intervention
Other: standard treatment — standard treatment according to EASL Clinical Practical Guidelines on the management of acute (fulminant) liver failure 2017.

SUMMARY:
Acute liver failure patients posed high mortality rate despite receiving standard therapy. The severity and mortality even higher in patients with underlying liver disease. Acute liver failure cause hyperinflammatory response in early stage and immunoparalysis in later stage. The surge of proinflammatory cytokines leads to multiorgan failure and more liver injury. Subsequent immunoparalysis may lead to lethal secondary infections.

Liver support system had been used in acute and acute ontop chronic liver disease for last several decades. Double plasma molecular adsorption system (DPMAS) is one of the promising non-biological liver support system that have been extensively investigated in acute ontop chronic liver failure from hepatits B viral. DPMAS circuit consist of BS330 (bilirubin adsorber) and HA330 (Cytokines adsorber). Thus, DPMAS can also remove various cytokines. The effect of DPMAS on immune function in these patients has not been explored.

Recent randomized controlled trial by Srisawat et al. demonstrated improvement of mHLA-DR in septic shock patients who received polymyxin B extracorporeal therapy compare to control arm. Since liver failure show change of immunological profile resemble to sepsis. Investigators proposed that removal of toxic liver toxins and lethal cytokines by DPMAS will improve immunological profiles in acute ontop chronic liver failure patients.

Investigators plan to conduct a randomized controlled trial in acute ontop chronic liver failure patients who admitted to intensive care unit. Investigators plan to compare the immunomodulatory effects of DPMAS with standard treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or more
2. Diagnosis of Acute ontop chronic liver failure by Asian Pacific association for the study of the liver (APASL) criteria
3. Admitted to intensive care unit

Exclusion Criteria:

1. Pregnancy
2. Received steroid treatment
3. Expected dead within 24 hour
4. WBC < 500/mm3
5. Allergy to DPMAS
6. History of organ transplant
7. Terminal illness with do not resuscitation order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
mHLA-DR expression | 7 days
  mHLA-DR expression

SECONDARY OUTCOMES:
survival rate | 28 days
  survival rate
Reduction of total bilirubin | 7 days
  Reduction of total bilirubin
hepatic encephalopathy grading | 28 days
  hepatic encephalopathy grading
subsequent bacterial infection | 28 days
  subsequent bacterial infection
CD11b expression | 7 days
  CD11b expression

CONTACTS AND LOCATIONS:
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided